CLINICAL TRIAL: NCT06835062
Title: The Effects of Clinical Pilates on Physical Fitness Parameters, Symptom Severity, and Kinesiophobia in Women With Premenstrual Syndrome.
Brief Title: Clinical Pilates' Impact on Fitness, Symptoms & Kinesiophobia in PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Meltem Kaya, Assistant Professor Meltem Kaya, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AtlasUmkaya04
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Premenstrual Syndrome; Pilates Exercise
Keywords: Premenstrual Syndrome; Physical Fitness; Kinesiophobia; Clinic Pilates
MeSH Terms: conditions — Premenstrual Syndrome; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pilates Group (Experimental)
  Interventions: Behavioral: Recommendations for Enhancing General Well-Being; Other: Clinical Pilates
- Control Group (Active Comparator)
  Interventions: Behavioral: Recommendations for Enhancing General Well-Being

INTERVENTIONS:
Behavioral: Recommendations for Enhancing General Well-Being — * Wear comfortable clothing and lie on your back. Place one hand on your abdomen. As you inhale through your nose, direct your breath towards your hand, and exhale through your mouth.
  * In the same position, place one hand on your abdomen, inhale through your nose, and expand your belly under your hand. As you exhale through your mouth, purse your lips and blow out the air from your lungs.
  * Engage in brisk walking at least three times a week.
  * Perform stretching exercises similar to yoga; try forward bends while standing and sitting.
  * Stay active throughout the month; you can dance, swim, or ride a bike.
  * Reduce your intake of tea and caffeine.
  * Increase your consumption of milk.
  * Drink plenty of water.
  * Reduce your intake of sugar-rich snacks such as chocolate.
  * Prioritize foods rich in calcium, as well as vitamins A, B, and E.
Other: Clinical Pilates — In addition to the general well-being recommendations, the Clinical Pilates Group participated in a total of 16 face-to-face, clinically based Pilates exercise training sessions over eight weeks, with two sessions per week, each lasting 50 minutes. The exercise training started at the end of the menstrual cycle.
  The clinical Pilates-based exercise program applied to the group was designed by the researcher. The number of repetitions, levels, and variations of the exercises were progressively adjusted by the researcher according to the participants' conditions.
  During the first session, the principles of clinical Pilates were explained, following the BASI Pilates method as described by Isacowitz. Participants were taught alignment, breathing, and core engagement techniques.
  Arms: Clinical Pilates Group

SUMMARY:
Premenstrual syndrome (PMS) is characterized by a series of somatic and psychological symptoms of varying severity that occur during the luteal phase of the menstrual cycle, affecting approximately 30% of women and resolving with menstruation. These symptoms impact daily activities, interpersonal relationships, social engagements, work efficiency, and educational productivity. PMS manifests with physical symptoms such as breast swelling and tenderness, fatigue, headaches, and weight gain, as well as psychological and emotional symptoms such as mood disorders, irritability, and stress. Symptoms typically subside with the onset of menstruation. There is no single accepted treatment for PMS. Due to conflicting findings in studies, various treatment methods are used, including lifestyle modifications, education, stress management techniques (such as massage, reflexology, and yoga), exercise, or medical support. Regular exercise is known to improve overall well-being. It prevents the decrease in endorphin secretion during the luteal phase of the menstrual cycle and has a positive impact on PMS symptoms, particularly mood disorders, fluid retention, and breast tenderness. Pilates-based exercise training is an approach that enhances muscle stability through effective, controlled movements while strengthening muscle groups associated with pain. Clinical Pilates-based exercise training is considered a preferable method for PMS management, as it is believed to improve functional capacity, pain management, mood disorders, endurance, flexibility, symptom severity, and fear of movement in individuals with PMS. Due to the limited number of studies in the literature on PMS, our study aims to investigate the effects of a clinical Pilates-based exercise program on functional fitness parameters, symptom severity, and kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* Having Premenstrual Syndrome (PMS)
* Being able to read and understand Turkish
* Willingness to participate in the study

Exclusion Criteria:

* Being in menopause or perimenopause
* Being pregnant
* Currently participating in or having engaged in a regular exercise program (other than clinical Pilates) within the past year
* Having comorbid orthopedic, musculoskeletal, psychological, or cardiovascular conditions that may affect test evaluations

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As the topic is premenstrual syndrome, the participant must have a menstrual cycle.
Enrollment: 40 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Body Composition (Waist Circumference) | 8 weeks
  -Waist Circumference: Measured in centimeters using a non-elastic measuring tape at the narrowest point between the lowest rib and the anterior superior iliac spine (ASIS). It was recorded in centimeters.
Body Composition (Hip Circumference) | 8 weeks
  -Hip Circumference: Measured in centimeters at the widest part of the gluteus maximus and at the level of the pubis using a measuring tape.
Body Composition (Waist-to-Hip Ratio) | 8 weeks
  It is calculated by dividing the circumference of the waist by the circumference of the hips.
Functional Capacity | 8 weeks
  To analyze the participants' functional capacity, the 6-Minute Walk Test (6MWT) was conducted in accordance with the American Thoracic Society (ATS) criteria.
  In this test, participants were instructed to walk at their own pace without running for six minutes along a 30-meter straight corridor. Standardized encouragement phrases were used throughout the test to maintain motivation.
  The test result was recorded as the total distance walked in meters.
Flexibility | 8 weeks
  The Sit and Reach Test is a simple and widely used test to measure the flexibility. For the measurement, a test bench was used with the following dimensions: 32 cm in height, 35 cm in length, and 45 cm in width. A 0-50 cm measurement ruler was placed on the upper surface of the bench, extending 15 cm beyond the edge where the participants' feet were positioned. Participants were seated on the floor with their bare feet extended straight towards the test bench. The measurement was taken at the farthest point reached, where they held the position for 2 seconds. Measure the distance reached in centimeters.
Endurance (Trunk Flexion Test) | 8 weeks
  The Trunk Flexion Endurance Test measures core muscle endurance, especially in the abdominals and lower back. The person sits with knees bent, leans back to 60 degrees, and holds the position as long as possible. The test stops when the person loses form or falls backward and records in seconds.
Endurance (Lateral Bridge Test) | 8 weeks
  The Lateral Bridge Test measures core and lateral trunk muscle endurance, especially the obliques. The person holds a side plank position with the body straight and hips lifted. The test ends when the hips drop or the person loses form and records in seconds..
Endurance (Modified Biering-Sorensen Test) | 8 weeks
  The Modified Biering-Sorensen Test measures endurance of the lower back extensor muscles. The person lies prone on a bench, with the upper body unsupported beyond the edge and legs secured. They hold a horizontal position for as long as possible. The test stops when the person can no longer maintain the position and records in seconds.
Endurance (Prone Bridge Test) | 8 weeks
  The Prone Bridge Test (Plank Endurance Test) measures core stability and endurance, focusing on the abdominals, lower back, and shoulders. The person holds a forearm plank position, keeping the body straight and avoiding sagging or lifting the hips. The test ends when the person can no longer maintain proper form and records in seconds.
Premenstrual Syndrome Scale | 8 weeks
  The Premenstrual Syndrome Scale consists of 44 questions and is a five-point Likert-type assessment tool with the following response options:
  1. - Never
  2. - Very little
  3. - Sometimes
  4. - Often
  5. - Always During the administration of the Premenstrual Syndrome Scale, participants were instructed to evaluate each item according to the period one week before menstruation, following the guidelines at the beginning of the scale. They were asked to mark the corresponding rating for each statement based on their experiences during this period.
Tampa Scale for Kinesiophobia | 8 weeks
  The Tampa Scale for Kinesiophobia is a 17-item questionnaire designed to measure the fear of movement and re-injury. It uses a 4-point Likert scale, with the following response options:
  1. - Strongly disagree
  2. - Disagree
  3. - Agree
  4. - Strongly agree
  A higher score on the scale indicates a greater level of kinesiophobia (fear of movement and re-injury).

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Kaya, Principal Investigator — Atlas University
Locations (2):
- Turkey (Türkiye) (2):
  - Atlas University, Istanbul
  - Istanbul Atlas University, Istanbul

IPD SHARING:
Plan to Share IPD: No